CLINICAL TRIAL: NCT03360110
Title: Clinical Validation Study of Phoebe Lens
Brief Title: Comparison of New Contact Lens With Current Marketed Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-17-60
Record Dates: First submitted 2017-11-21; First posted 2017-12-02 (Actual); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double masked (participant, investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test lens (Active Comparator): Subjects randomized to wear pair of test lens either first or second
  Interventions: Device: Phoebe test lens; Device: stenfilcon A lens (control)
- stenfilcon A lens (control) (Active Comparator): Subjects randomized to wear pair of control lens either first or second
  Interventions: Device: Phoebe test lens; Device: stenfilcon A lens (control)

INTERVENTIONS:
Device: Phoebe test lens — Daily disposable contact lens
  Other Names: Test Lens; Phoebe Contact Lens
Device: stenfilcon A lens (control) — Daily disposable contact lens
  Other Names: MyDay daily disposable contact lens

SUMMARY:
The purpose of this study is to validate the clinical performance of a new contact lens design.

DETAILED DESCRIPTION:
Evaluate the clinical performance of its Phoebe contact lenses (Test) compared to the commercially available MyDay contact lenses (Control).

ELIGIBILITY:
Inclusion criteria

A person is eligible for inclusion in the study if he/she:

* Between and 18 and 35 years of age and has full legal capacity to volunteer
* Has had a self-reported oculo-visual examination in the last two years
* Has read and understood the information consent letter
* Is willing and able to follow instructions and maintain the appointment schedule
* Is correctable to a visual acuity of 20/25 or better (in each eye) with their habitual correction or 20/20 best corrected
* Has a Contact Lens Refraction between -1.00D and -6.00D
* Cylinder power ≤ -0.75DC in Spherical Cylindrical Refraction
* Currently wears soft contact lenses
* Is willing to wear lenses for a minimal of 8 hours a day and everyday during the course of the study
* Has clear corneas and no active ocular disease
* Has not worn lenses for at least 12 hours before the first visit

Exclusion Criteria

A person will be excluded from the study if he/she:

* Has never worn contact lenses before
* Is wearing Monovision modality
* Has any systemic disease affecting ocular health
* Is using any systemic or topical medications that will affect ocular health
* Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye
* Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars
* Is aphakic
* Has undergone corneal refractive surgery
* Is participating in any other type of eye related clinical or research study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Kolbaum, O.D., Ph.D., FAAO, FBCLA, Principal Investigator — Clinical Optics Research Lab (CORL), Indiana University
Locations (1):
- Clinical Optical Research Lab (CORL), Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Lens, Then Control Lens: Subjects randomized to wear pair of test lens, then control lens. Each lens type was worn for three days using a daily wear / daily replacement schedule.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
- Control Lens, Then Test Lens: Subjects randomized to wear pair of control lens, then test lens. Each lens type was worn for three days using a daily wear / daily replacement schedule.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
Period: First Intervention
Arm/Group | Test Lens, Then Control Lens | Control Lens, Then Test Lens
Started | 27 | 26
Completed | 27 | 26
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Test Lens, Then Control Lens | Control Lens, Then Test Lens
Started | 27 | 26
Completed | 27 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were six (6) protocol deviations and data was not included in the analyses.
Groups:
- Overall Study: Subjects randomized to wear pair of test/control lens either first or second, then wear other lens.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
Arm/Group | Overall Study
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 47
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Corneal Staining Extent
Description: Measurement of extent of corneal staining using Fluorescein, blue light, yellow filter, full beam, medium magnification on a scale 0-4 (0=no staining, 1 = 1-15% of area, 2= 16-30% of area, 3=31-45% of area, 4=>45% of area).
Time Frame: Baseline
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Phoebe Test Lens: Subjects randomized to wear pair of test lens, then control lens. Each lens type was worn for three days using a daily wear / daily replacement schedule.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
- Stenfilcon A Control Lens: Subjects randomized to wear pair of control lens, then test lens. Each lens type was worn for three days using a daily wear / daily replacement schedule.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
Arm/Group | Phoebe Test Lens | Stenfilcon A Control Lens
Number analyzed (Participants) | 47 | 47
Number analyzed (Eyes) | 94 | 94
units on a scale | 0.04 (0.09) | 0.04 (0.09)

2. Primary Outcome: Corneal Staining Extent
Description: as for outcome 1
Time Frame: Day 3
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Phoebe Test Lens | Stenfilcon A Control Lens
Number analyzed (Participants) | 47 | 47
Number analyzed (Eyes) | 94 | 94
units on a scale | 0.07 (0.13) | 0.07 (0.12)

3. Primary Outcome: Conjunctival Staining Score
Description: Amount of staining observed on the conjunctiva scored 0-4 (0=none, 4=Deep Confluent, in 0.50 steps
Time Frame: Baseline
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Phoebe Test Lens | Stenfilcon A Control Lens
Number analyzed (Participants) | 47 | 47
Number analyzed (Eyes) | 94 | 94
score on a scale | 0.18 (0.21) | 0.18 (0.21)

4. Primary Outcome: Conjunctival Staining Score
Description: Amount of staining observed on the conjunctiva scored 0-4 (0=none, 4=Deep Confluent, in 0.50 steps
Time Frame: Day 3
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Phoebe Test Lens | Stenfilcon A Control Lens
Number analyzed (Participants) | 47 | 47
Number analyzed (Eyes) | 94 | 94
score on a scale | 0.26 (0.26) | 0.29 (0.28)

5. Primary Outcome: Palpebral Hyperemia on Upper Lid
Description: Measurement of hyperemia of the palpebral conjunctiva; graded 0-4 (0=none, 4=severe) in 0.25 steps
Time Frame: Baseline
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Phoebe Test Lens: Upper Lid: Subjects randomized to wear pair of test lens, then control lens. Each lens type was worn for three days using a daily wear / daily replacement schedule. Upper lid was assessed for palpebral hyperemia.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
- Stenfilcon A Control Lens: Upper Lid: Subjects randomized to wear pair of control lens, then test lens. Each lens type was worn for three days using a daily wear / daily replacement schedule. Upper lid was assessed for palpebral hyperemia.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
Arm/Group | Phoebe Test Lens: Upper Lid | Stenfilcon A Control Lens: Upper Lid
Number analyzed (Participants) | 47 | 47
Number analyzed (Eyes) | 94 | 94
units on a scale | 0.96 (0.39) | 0.96 (0.39)

6. Primary Outcome: Palpebral Hyperemia on Upper Lid
Description: Measurement of hyperemia of the palpebral conjunctiva; graded 0-4 (0=none, 4=severe) in 0.25 steps
Time Frame: Day 3
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Phoebe Test Lens: Upper Lid | Stenfilcon A Control Lens: Upper Lid
Number analyzed (Participants) | 47 | 47
Number analyzed (Eyes) | 94 | 94
units on a scale | 1.05 (0.40) | 1.06 (0.38)

7. Primary Outcome: Palpebral Hyperemia on Lower Lid
Description: Measurement of hyperemia of the palpebral conjunctiva; graded 0-4 (0=none, 4=severe) in 0.25 steps
Time Frame: Baseline
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Phoebe Test Lens: Lower Lid: Subjects randomized to wear pair of test lens, then control lens. Each lens type was worn for three days using a daily wear / daily replacement schedule. Lower lid was assessed for palpebral hyperemia.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
- Stenfilcon A Control Lens: Lower Lid: Subjects randomized to wear pair of control lens, then test lens. Each lens type was worn for three days using a daily wear / daily replacement schedule. Lower lid was assessed for palpebral hyperemia.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
Arm/Group | Phoebe Test Lens: Lower Lid | Stenfilcon A Control Lens: Lower Lid
Number analyzed (Participants) | 47 | 47
Number analyzed (Eyes) | 94 | 94
units on a scale | 0.96 (0.39) | 0.96 (0.39)

8. Primary Outcome: Palpebral Hyperemia on Lower Lid
Description: Measurement of hyperemia of the palpebral conjunctiva; graded 0-4 (0=none, 4=severe) in 0.25 steps
Time Frame: Day 3
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Phoebe Test Lens: Lower Lid | Stenfilcon A Control Lens: Lower Lid
Number analyzed (Participants) | 47 | 47
Number analyzed (Eyes) | 94 | 94
units on a scale | 1.05 (0.40) | 1.06 (0.38)

9. Primary Outcome: Palpebral Roughness Grade - Upper Lid
Description: Measurement of smoothness of palpebral conjunctiva; graded 0-4 (0=smooth, 4=severe) in 0.25 steps
Time Frame: Baseline
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Phoebe Test Lens: Upper Lid: Subjects randomized to wear pair of test lens, then control lens. Each lens type was worn for three days using a daily wear / daily replacement schedule. Upper lid was assessed for palpebral roughness.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
- Stenfilcon A Control Lens: Upper Lid: Subjects randomized to wear pair of control lens, then test lens. Each lens type was worn for three days using a daily wear / daily replacement schedule. Upper lid was assessed for palpebral roughness.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
Arm/Group | Phoebe Test Lens: Upper Lid | Stenfilcon A Control Lens: Upper Lid
Number analyzed (Participants) | 47 | 47
Number analyzed (Eyes) | 94 | 94
units on a scale | 1.09 (0.51) | 1.09 (0.51)

10. Primary Outcome: Palpebral Roughness Grade - Upper Lid
Description: Measurement of smoothness of palpebral conjunctiva; graded 0-4 (0=smooth, 4=severe) in 0.25 steps
Time Frame: Day 3
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Phoebe Test Lens: Upper Lid | Stenfilcon A Control Lens: Upper Lid
Number analyzed (Participants) | 47 | 47
Number analyzed (Eyes) | 94 | 94
units on a scale | 1.26 (0.53) | 1.20 (0.46)

11. Primary Outcome: Palpebral Roughness Grade - Lower Lid
Description: Measurement of smoothness of palpebral conjunctiva; graded 0-4 (0=smooth, 4=severe) in 0.25 steps
Time Frame: Baseline
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Phoebe Test Lens: Lower Lid: Subjects randomized to wear pair of test lens, then control lens. Each lens type was worn for three days using a daily wear / daily replacement schedule. Lower lid was assessed for palpebral roughness.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
- Stenfilcon A Control Lens: Lower Lid: Subjects randomized to wear pair of control lens, then test lens. Each lens type was worn for three days using a daily wear / daily replacement schedule. Lower lid was assessed for palpebral roughness.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
Arm/Group | Phoebe Test Lens: Lower Lid | Stenfilcon A Control Lens: Lower Lid
Number analyzed (Participants) | 47 | 47
Number analyzed (Eyes) | 94 | 94
units on a scale | 1.07 (0.50) | 1.07 (0.50)

12. Primary Outcome: Palpebral Roughness Grade - Lower Lid
Description: Measurement of smoothness of palpebral conjunctiva; graded 0-4 (0=smooth, 4=severe) in 0.25 steps
Time Frame: Day 3
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Phoebe Test Lens: Lower Lid | Stenfilcon A Control Lens: Lower Lid
Number analyzed (Participants) | 47 | 47
Number analyzed (Eyes) | 94 | 94
units on a scale | 1.23 (0.52) | 1.20 (0.46)

13. Secondary Outcome: Distance Visual Acuity
Description: Distance visual acuity recorded in logMAR.
Time Frame: Baseline (at lens dispense)
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: Log(MAR)
Groups:
- Phoebe Test Lens: Dispense: Subjects randomized to wear pair of test lens, then control lens. Each lens type was worn for three days using a daily wear / daily replacement schedule.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
- Stenfilcon A Control Lens: Dispense: Subjects randomized to wear pair of control lens, then test lens. Each lens type was worn for three days using a daily wear / daily replacement schedule.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
Arm/Group | Phoebe Test Lens: Dispense | Stenfilcon A Control Lens: Dispense
Number analyzed (Participants) | 47 | 47
Log(MAR)
  High Illumination High Contrast, Binocular | -0.23 (0.06) | -0.22 (0.06)
  Low Illumination High Contrast, Binocular | -0.03 (0.08) | -0.03 (0.07)

14. Secondary Outcome: Distance Visual Acuity
Description: Distance visual acuity recorded in logMAR.
Time Frame: Day 3
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: Log(MAR)
Groups:
- Phoebe Test Lens: 3 Days: Subjects randomized to wear pair of test lens, then control lens. Each lens type was worn for three days using a daily wear / daily replacement schedule.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
- Stenfilcon A Control Lens: 3 Days: Subjects randomized to wear pair of control lens, then test lens. Each lens type was worn for three days using a daily wear / daily replacement schedule.
  Phoebe test lens: Daily disposable contact lens
  stenfilcon A lens (control): Daily disposable contact lens
Arm/Group | Phoebe Test Lens: 3 Days | Stenfilcon A Control Lens: 3 Days
Number analyzed (Participants) | 47 | 47
Log(MAR)
  High Illumination High Contrast, Binocular | -0.23 (0.06) | -0.22 (0.06)
  Low Illumination High Contrast, Binocular | -0.04 (0.06) | -0.04 (0.07)

15. Secondary Outcome: Near Visual Acuity
Description: Near visual acuity recorded in logMAR
Time Frame: Baseline (at dispense)
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: Log(MAR)
Arm/Group | Phoebe Test Lens: Dispense | Stenfilcon A Control Lens: Dispense
Number analyzed (Participants) | 47 | 47
Log(MAR)
  High Illumination High Contrast, Binocular | -0.16 (0.07) | -0.16 (0.06)
  Low Illumination High Contrast, Binocular | 0.09 (0.10) | 0.06 (0.09)

16. Secondary Outcome: Near Visual Acuity
Description: Near visual acuity recorded in logMAR
Time Frame: Day 3
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: Log(MAR)
Arm/Group | Phoebe Test Lens: 3 Days | Stenfilcon A Control Lens: 3 Days
Number analyzed (Participants) | 47 | 47
Log(MAR)
  High Illumination High Contrast, Binocular | -0.17 (0.07) | -0.19 (0.07)
  Low Illumination High Contrast, Binocular | 0.06 (0.09) | 0.04 (0.09)

17. Secondary Outcome: Vision Quality Rating
Description: Subjective vision quality rated on a 0-10 scale (0=extremely poor, 10=excellent)
Time Frame: Baseline (at dispense)
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phoebe Test Lens | Stenfilcon A Control Lens
Number analyzed (Participants) | 47 | 47
units on a scale | 9.2 (1.0) | 9.3 (0.07)

18. Secondary Outcome: Vision Quality Rating
Description: Subjective vision quality rated on a 0-10 scale (0=extremely poor, 10=excellent)
Time Frame: Day 3
Population: There were 6 protocol deviations reported in this study and data from the 6 subjects were not used for data analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phoebe Test Lens | Stenfilcon A Control Lens
Number analyzed (Participants) | 47 | 47
units on a scale | 9.3 (0.9) | 9.2 (1.0)

ADVERSE EVENTS:
Time Frame: From dispense up to three days for each intervention.
Groups:
- Test Lens: Subjects were randomized to wear pair of test lens for 3 days.
  Phoebe test lens: Daily disposable contact lens
- Stenfilcon A Lens (Control): Subjects were randomized to wear pair of control lens for 3 days.
  stenfilcon A lens (control): Daily disposable contact lens
Arm/Group | Test Lens | Stenfilcon A Lens (Control)
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT03360110/Prot_SAP_000.pdf